CLINICAL TRIAL: NCT03335501
Title: An Open-label, Double-blind, Randomized, Two-way, Cross-over Pilot Study to Provide Preliminary Evidence of the Efficacy of Rapid-acting Aspart Compared to Faster Acting Aspart Within the Context of Single-hormone Closed-loop Strategy at Regulating Postprandial Glucose Levels in Adults With Type 1 Diabetes
Brief Title: Comparison of the Efficacy of Rapid-acting Aspart and Faster Acting Aspart Within the Context of Single-hormone Closed-loop Strategy at Regulating Postprandial Glucose Levels
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The owner of the algorithm does not wish that this study be undertaken
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLASS-FiAsp
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Closed-loop control; Artificial pancreas; Postprandial glucose control; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Infusion Systems; Continuous Glucose Monitoring; Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid-acting Aspart (Active Comparator): Rapid-acting Aspart will be used to regulate glucose levels
  Interventions: Device: Insulin pump; Device: Continuous glucose monitoring system; Other: 11-hour intervention with the single-hormone artificial pancreas
- Faster insulin Aspart (Active Comparator): Faster insulin Aspart will be used to regulate glucose levels
  Interventions: Device: Insulin pump; Device: Continuous glucose monitoring system; Other: 11-hour intervention with the single-hormone artificial pancreas

INTERVENTIONS:
Device: Insulin pump — The participant's insulin pump will be used to infuse insulin
Device: Continuous glucose monitoring system — The Dexcom G4 Platinum will be used to measure glucose levels
Other: 11-hour intervention with the single-hormone artificial pancreas — Subjects will be admitted at IRCM at 9:30. An intravenous catheter will be inserted into an arm or a hand vein for blood sampling purposes. A cartridge containing rapid-acting Aspart or faster acting Aspart will be placed in the insulin pump. Closed-loop strategy will start at 10:00 until 21:00. A glucose sensor reading will be entered manually into the computer every 10 minutes. The computer will generate a recommendation for the basal rates of insulin delivery. Pumps' parameters will then be changed manually to implement the computer generated recommendations.
  At 12:00, a lunch meal will be served. An insulin bolus will be given 15 minutes before the meal. At 17:00, a dinner meal will be served. As recommended, an insulin bolus will be given at the time of the meal. Each subject will ingest the same meals during both visits.
  Venous blood samples will be obtained for the measurement of plasma glucose and insulin concentrations. Blood samples will be taken every 20 minutes.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings.

The objective of this pilot study is to inform both the decision whether to conduct a confirmatory study and the design of the larger confirmatory trial. In addition, we want to estimate postprandial glucose levels parameters and confidence interval in an 11-hour in-patient study with standardized conditions in adults with type 1 diabetes, estimate the size and direction of the treatment effect.

Faster insulin Aspart (FiAsp) will provide preliminary evidence of efficacy to regulate postprandial glucose levels compared to rapid-acting Aspart in adults with type 1 diabetes using insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 6 months.
4. HbA1c ≤ 12%.

Exclusion Criteria:

1. Using a patch-pump (e.g. Omnipod)
2. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
3. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
4. Ongoing or planned pregnancy.
5. Breastfeeding.
6. Severe hypoglycemic episode within two weeks of screening.
7. Current use of glucocorticoid medication (except low stable dose and inhaled stable treatment).
8. Known or suspected allergy to the trial products or meal contents.
9. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
10. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc).
11. Problems with venous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glucose levels 1 hour after the meal | 1 hour

SECONDARY OUTCOMES:
Area under the curve of plasma glucose levels for the 1-hour period following the meal. | 1 hour
Area under the curve of plasma glucose levels for the 2-hour period following the meal. | 2 hours
Plasma glucose level 1 hour after the meal. | 1 hour
Plasma glucose level 2 hours after the meal. | 2 hours
Glycemic peak in the 3 hours following the meal. | 3 hours
Change in plasma glucose levels 2 hours after the meal. | 2 hours
Peak time of glucose levels over the 4 hours following the meal. | 4 hours
Number of hypoglycemic events less than 4.0 mmol/L over the 4 hours following the meal. | 4 hours
Percentage of time of plasma glucose levels between 3.9 and 7.8 mmol/L. | 11 hours
Percentage of time of sensor glucose levels between 3.9 and 7.8 mmol/L. | 11 hours
Percentage of time of plasma glucose levels between 3.9 and 10 mmol/L. | 11 hours
Percentage of time of sensor glucose levels between 3.9 and 10 mmol/L. | 11 hours
Percentage of time of plasma glucose levels below 3.9 mmol/L. | 11 hours
Percentage of time of sensor glucose levels below 3.9 mmol/L. | 11 hours
Percentage of time of plasma glucose levels below 3.3 mmol/L. | 11 hours
Percentage of time of sensor glucose levels below 3.3 mmol/L. | 11 hours
Percentage of time of plasma glucose levels below 2.8 mmol/L. | 11 hours
Percentage of time of sensor glucose levels below 2.8 mmol/L. | 11 hours
Percentage of time of plasma glucose levels above 10 mmol/L. | 11 hours
Percentage of time of sensor glucose levels above 10 mmol/L. | 11 hours
Percentage of time of plasma glucose levels above 13.9 mmol/L | 11 hours
Percentage of time of sensor glucose levels above 13.9 mmol/L | 11 hours
Percentage of time of plasma glucose levels above 16.7 mmol/L. | 11 hours
Percentage of time of sensor glucose levels above 16.7 mmol/L. | 11 hours
Area under the curve of plasma glucose levels below 3.9 mmol/L. | 11 hours
Area under the curve of sensor glucose levels below 3.9 mmol/L. | 11 hours
Area under the curve of plasma glucose levels below 3.3 mmol/L. | 11 hours
Area under the curve of sensor glucose levels below 3.3 mmol/L. | 11 hours
Area under the curve of plasma glucose levels below 2.8 mmol/L. | 11 hours
Area under the curve of sensor glucose levels below 2.8 mmol/L. | 11 hours
Area under the curve of plasma glucose levels above 10.0 mmol/L. | 11 hours
Area under the curve of sensor glucose levels above 10.0 mmol/L. | 11 hours
Area under the curve of plasma glucose levels above 13.9 mmol/L. | 11 hours
Area under the curve of sensor glucose levels above 13.9 mmol/L. | 11 hours
Area under the curve of plasma glucose levels above 16.7 mmol/L. | 11 hours
Area under the curve of sensor glucose levels above 16.7 mmol/L. | 11 hours
Standard deviation of plasma glucose levels. | 11 hours
Standard deviation of sensor glucose levels. | 11 hours
Coefficient of variance of plasma glucose levels. | 11 hours
Coefficient of variance of sensor glucose levels. | 11 hours
Total insulin delivery. | 11 hours
Mean plasma glucose level. | 11 hours
Mean sensor glucose level. | 11 hours
Mean plasma insulin concentration. | 11 hours
Number of hypoglycemic events less than 3.3 mmol/L (>20 minutes). | 11 hours

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal